CLINICAL TRIAL: NCT06739239
Title: French COhoRte Extra-Vascular Implantable CardiovErter DefibrillatoR
Acronym: FOREVER
Status: Recruiting | Type: Observational
Sponsor: Paris Sudden Death Expertise Center (Other)
Collaborators: European Georges Pompidou Hospital (Other); University Hospital, Grenoble (Other); University Hospital, Clermont-Ferrand (Other); University Hospital, Rouen (Other); Centre Hospitalier Universitaire de Besancon (Other); Clinique du Millenaire (Other); Institut Mutualiste Montsouris (Other); Groupe Hospitalier Pitie-Salpetriere (Other); University Hospital, Lille (Other); University Hospital, Caen (Other); Hospices Civils de Lyon (Other); CHU de la Timone, Marseille, France (Unknown); Centre Cardio-Thoracique de Monaco (Unknown); Hospital of Lens (Unknown); Institute Arnault Tzanck, France (Other); University Hospital, Strasbourg, France (Other); University Hospital, Limoges (Other); University Hospital, Montpellier (Other); Clinique Pasteur Toulouse (Other); University Hospital, Bordeaux (Other); University Hospital, Toulouse (Other); Institut Jacques Cartier - Massy (Unknown); Clinique Saint Augustin - Bordeaux (Unknown); Rennes University Hospital (Other); Clinique de la Sauvegarde (Other); University Hospital of Saint-Etienne (Other); Centre Hospitalier Universitaire, Amiens (Other); Poitiers University Hospital (Other); Clinique Saint-Gatien - Tours (Unknown); CHU de Reims (Other); Centre Hospitalier Universitaire Dijon (Other); Hospital St. Joseph, Marseille, France (Other); Centre Hospitalier Annecy Genevois (Other); Clinique St Pierre, Perpignan, France (Unknown); Bichat Hospital (Other); Universite de La Reunion (Other); University Hospital Center of Martinique (Other); Henri Mondor University Hospital (Other); University Hospital, Angers (Other Government); Central Hospital, Nancy, France (Other); Hôpital privé Clairval - Marseille (Unknown); Médipôle Lyon-Villeurbanne (Other); Hôpital Privé Les Franciscaines (Other); Hospital Ambroise Paré Paris (Other); Central Hospital, Metz Thionville, France (Unknown); Hopital Prive Saint Martin - Bordeaux (Unknown); Hôpital Privé de Parly II - Le Chesnay (Other)
Responsible Party: Principal Investigator, Marijon, Head of Cardiology Division, European Georges Pompidou Hospital
Other Study IDs: 2236443v0
Record Dates: First submitted 2024-12-01; First posted 2024-12-18 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Defibrillators, Implantable; Sudden Cardiac Death Due to Cardiac Arrhythmia
Keywords: Implantable cardioverter defibrillator; sudden cardiac death; Extravascular Implantable Cardioverter-Defibrillator
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- All patients implanted with EV-ICD in France
  Interventions: Device: Extra-Vascular Implantable Cardioverter Defibrillator

INTERVENTIONS:
Device: Extra-Vascular Implantable Cardioverter Defibrillator — The pulse generator is implanted along the patient's left midaxillary line, and the lead is positioned substernally.

SUMMARY:
Implantable cardioverter-defibrillators (ICDs) are widely recognized for their efficacy in reducing the risk of sudden cardiac death in high-risk patients. Nonetheless, there remains significant scope for improving outcomes through advancements in device technology and design. The extravascular cardioverter-defibrillator (EV-ICD) represents such an innovation, offering key advantages over other ICD systems. It incorporates a lead positioned in the substernal space, enabling the delivery of pause-prevention security pacing, antitachycardia pacing, and defibrillation energy similar to that provided by conventional transvenous ICDs.

Previous studies have demonstrated that EV-ICDs can be implanted safely and are capable of terminating majority of induced ventricular arrhythmias during implantation; however, follow-up data are limited to highly experienced selected centers and over a relatively small follow-up period (6-month follow-up). The FOREVER cohort study, initiated by the French Institute of Health and Medical Research, aims to evaluate the EV-ICD use in France.

This nationwide evaluation will provide an exhaustive collection of all EV-ICD implantations in France, offering valuable real-world evidence on the long-term safety and efficacy of the device.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing EV-ICD implantation

Exclusion Criteria:

* Refusal of consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients implanted with an EV-ICD in France.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Appropriate Therapies | Through the study completion, an average of 5 years
  The incidence of ICD shocks or ICD ATPs.
EV-ICD-related Early Complications (Prior to Hospital Discharge) | Through the study completion, an average of 5 years
  The incidence of each complication related to the procedure or the device: pocket hematoma, infection, poor wound healing, inappropriate shocks, lead issues, pneumothorax, pericardial injury, other complications with details.
EV-ICD related Late Complications (After Hospital Discharge) | Through the study completion, an average of 5 years
  The incidence of each complication related to the device or genetaor change procedure: infection, pocket hematoma, poor wound healing, inappropriate shocks, lead issues, premature battery depletion, chronic pain, painful pacing, EV-ICD related death
Overall and Specific Mortalities | Through the study completion, an average of 5 years
  Incidence of deaths. Causes of Deaths: cardiovascular cause with the main raison leading to death, non-cardiovascular cause with the main raison leading to death, EV-ICD related death with details, and unknown cause.

SECONDARY OUTCOMES:
Interventions During Follow-up | Through the study completion, an average of 5 years
  Incidence and type of all EV-ICD related intervention. Raison of reintervention: complication, type of complication, generator change and pacing need.
Heart Transplantation | Through the study completion, an average of 5 years
  The incidence of heart transplant during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- European Georges Pompidou Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data (IPD) related to the primary and secondary outcomes of the study will be made available. This includes baseline characteristics, procedural details, follow-up outcomes, and information on complications or adverse events. All shared data will exclude any information that could potentially identify participants.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: From 01/01/2030 to 01/01/2035
Access Criteria: Access to the data will be granted upon reasonable request from qualified researchers, with active involvement of the study team in the project.